CLINICAL TRIAL: NCT04233619
Title: Correlation of Microvascular Ophthalmic Disease With Macrovascular Coronary Artery Disease in Trinidad: The EYE-MI TNT Study
Brief Title: Correlation of Microvascular Ophthalmic Disease With Macrovascular Coronary Artery Disease in Trinidad
Acronym: EYE-MI TNT
Status: Completed | Type: Observational
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Other Study IDs: CEC819/01/19
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2021-02

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: optical coherence tomography — non-invasive test performed by an Ophthalmologist that allows three-dimensional imaging of the retinal vasculature

SUMMARY:
Coronary artery disease (CAD) is the leading cause of death in Trinidad and Tobago. Early detection and management can help improve morbidity and mortality. Retinal artery microvascular disease has been shown to directly correlate with coronary artery disease. Retinal artery calibre screening via the Optic Coherence Tomography (OCT) will provide a non-invasive method of diagnosing CAD.

DETAILED DESCRIPTION:
Cardiovascular disease is the number one cause of death in Trinidad and Tobago. There has been a 20.4% increase in cardiovascular deaths from 2007 to 2017(1). Prevention of non-communicable diseases decreases the burden and progression to cardiovascular disease. Prevention of death from cardiovascular disease can also be decreased by early detection, intervention and appropriate management of coronary artery disease.

Due to the burden of the cost of health care on the economy of Trinidad and Tobago, patients are required to go on a waitlist to receive specialist medical investigation such as a coronary angiogram. This investigation is only offered at one public health facility in Trinidad and Tobago, the Eric Williams Medical Sciences Complex.

Coronary artery disease is graded by a scoring system, the SYNTAX score, which is calculated based on the assessment of the complexity of coronary artery disease by coronary angiography (2). In a study done on 173 patients- the EYE-MI study, patients with the lowest retinal vascular density had a higher SYNTAX score, indicating a direct correlation between retinal artery calibre and the severity of coronary artery disease (3).

Retinal artery calibre is assessed using the Optical Coherence Tomography. It is a relatively affordable non-invasive test performed by an Ophthalmologist that allows three dimensional imaging of the retinal vasculature. It is recommended by the American Association of Ophthalmologist for assessing retinal disease (4). This test is not available in the public health care system in Trinidad and Tobago.

In a country with a Human Capital Index of 0.61 (5), and cardiovascular disease being the number one cause of death, a cheaper non-invasive tool to screen for coronary artery disease would be of benefit to the population. We postulate that there is a direct correlation between the retinal artery calibre assessed by the Optical Coherence Tomography and the severity of coronary artery disease. There are not many studies assessing this relationship and this study will promote further avenues for research into this correlation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and over,
2. Patients who had a coronary angiogram done at the Catheterisation lab at the Eric Williams Medical Sciences Complex during the study period.

Exclusion Criteria:

1. Patients who do not give informed consent to participate in the study,
2. Patients who are acutely unwell,
3. Patients who are symptomatic for Coronary Artery Disease,
4. Patients with bilateral cataract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both male and female gender; all racial/ethnic groups including Afro-Caribbean, Indo-Caribbean, Asians, Caucasians, Hispanics and mixed ethnicities will be included in the study. Potential subjects will be identified from the Catheterization Lab at the Eric Williams Medical Sciences Complex. Patients who underwent or undergoing coronary angiography at the Eric Williams Medical Sciences Complex from May 1st 2019 to April 30th 2021.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
To determine if there is a direct correlation between retinal artery calibre and coronary artery disease | 2 years
  Compare SYNTAX score and OCT results to determine correlation

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Saint Augustine, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yammine M, Itagaki S, Pawale A, Toyoda N, Reddy RC. SYNTAX score may predict the severity of atherosclerosis of the ascending aorta. J Thorac Dis. 2017 Oct;9(10):3859-3865. doi: 10.21037/jtd.2017.09.17. PMID 29268395
- [Background] Michelson EL, Morganroth J, Nichols CW, MacVaugh H 3rd. Retinal arteriolar changes as an indicator of coronary artery disease. Arch Intern Med. 1979 Oct;139(10):1139-41. PMID 485746
- [Derived] Seecheran NA, Rafeeq S, Maharaj N, Swarath S, Seecheran V, Seecheran R, Seebalack V, Jagdeo CL, Seemongal-Dass R, Quert AYL, Giddings S, Ramlackhansingh A, Sandy S, Motilal S, Seemongal-Dass R. Correlation of RETINAL Artery Diameter with Coronary Artery Disease: The RETINA CAD Pilot Study-Are the Eyes the Windows to the Heart? Cardiol Ther. 2023 Sep;12(3):499-509. doi: 10.1007/s40119-023-00320-x. Epub 2023 Jun 15. PMID 37318673